CLINICAL TRIAL: NCT06624657
Title: Concurrent Effects of High-intensity Interval Training and Vitamin D Supplementation on Bone Metabolism Among Women Diagnosed With Osteoporosis
Brief Title: High-intensity Interval Training and Vitamin D Effects on Bone Metabolism Among Women Diagnosed With Osteoporosis
Status: Completed | Type: Observational
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Sami Gabr, King Saud University, King Saud University
Other Study IDs: RRC-2016-028
Record Dates: First submitted 2024-09-29; First posted 2024-10-03 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis; Exercise Overtraining; Vitamin D 25-Hydroxylase Deficiency
Keywords: Exercise training, BMD, osteoporosis, Vitamin D deficiency
MeSH Terms: conditions — Osteoporosis; Overtraining Syndrome; Vitamin D Hydroxylation-Deficient Rickets, Type 1B; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Height, weight, BMI measurements, Serum levels of vitamin 25(OH) D, osteocalcin, s-BAP, and calcium ,and, BMD of the lumbar spine (L2-L4) and hip were identified in subjects of all groups pre ad post HIIT and vitamin D supplementation for 16 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- control group: Participants are women with osteoporosis Characterized by normal daily activities and diets
  Interventions: Other: vitamin D supplements fo 16 weks
- Exercise group: Participants are women's with osteoporosis participated in HIIT-exercise program interventions for 16 weeks
  Interventions: Other: vitamin D supplements fo 16 weks
- Vitamin D group: Participants are women's with osteoporosis who received vitamin D 800IU/ day for 16 weeks
  Interventions: Other: vitamin D supplements fo 16 weks
- Concurrent group: Participants are women's with osteoporosis who shared for HIIT exercise program plus vitamin D for 16 weeks
  Interventions: Other: vitamin D supplements fo 16 weks

INTERVENTIONS:
Other: vitamin D supplements fo 16 weks — subjects exercised by HIIT-exercise for 16 weeks
  Other Names: HIIT-exercise for 16 weeks

SUMMARY:
The effects of 16-week high-intensity interval training (HIIT) and vitamin D supplements on bone mineral density (BMD) in women with osteoporosis. The participants assigned for HITT exercise training with or without vitamin D supplements for 16 weeks, and the levels of serum bone parameters like, Osteocalcin (OC), Ca, and s-BAP were estimated in women with osteoporosis at baseline and after post-training interventions. In addition, the levels of Vitamin D were also identified in all women's accordingly.

DETAILED DESCRIPTION:
our study aimed to investigate the effects of 16-week high-intensity interval training (HIIT) and vitamin D supplements on bone mineral density (BMD) in women with osteoporosis. thus, Serum levels of 25-Hydroxy-vitamin D (OH-D), Osteocalcin (OC), Ca, and s-BAP were estimated in women with osteoporosis at baseline and after post-training interventions. One-hundred twenty sedentary women aged (30-50 years) were diagnosed with osteoporosis. Patients were classified into four groups, 30 patients in each group; Control group (normal daily activities); Exercise group (HIIT-exercise for 16 weeks); Vitamin D group (vitamin D 800IU/ day for 16 weeks), and Concurrent group (HIIT exercise plus vitamin D for 16 weeks). Anthropometric measurements, BMD, serum levels of vitamin 25-(OH) D, Osteocalcin, s-BAP, and calcium were estimated in all participants' pre- and post-exercise training.

ELIGIBILITY:
Inclusion Criteria:

* A healthy non-smoker premenopausal women's
* Age are 30-50 years old
* subjects who diagnosed with osteoporosis based on the clinical features of bone mineral density (BMD) measured from both lumbar spine L2 to L4, and from the right and left sides of the hip region by Dual Energy X-ray Absorptiometry (DEXA, UNIGAMMA PLUS AC 230V 50/60Hz 400w, USA) scan method.

Exclusion Criteria:

* Women with; physical disability,
* abnormal hormonal levels
* severe disease complications such as chronic kidney and liver diseases,
* rheumatoid and osteoarthritis diseases
* significant overweight (BMI ≥25) and obesity (≥30 kg/m2) per recommended by the World Health Organization
* history of receiving calcium, multivitamin supplements, corticosteroids, anticonvulsants, and heparin which might affects up on the assessment of bone markers and BMD measurements were excluded from this study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: a healthy, no-smoking premenopausal women aged (30-50) years old subjects who diagnosed with osteoporosis based on the clinical features and diagnosis evidence of bone mineral density (BMD) measured from both lumbar spine L2 to L4, and from the right and left sides of the hip region by Dual Energy X-ray Absorptiometry (DEXA, UNIGAMMA PLUS AC 230V 50/60Hz 400w, USA) scan method were invited to participate in this study
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurements | 4 month
  BMI measurements were evaluated

SECONDARY OUTCOMES:
Assessments of bone mineral density (BMD) | 4 month
  Before and after training along with vitamin D supplements, BMD of the lumbar spine
Assessments of bone serum markers and vitamin 25(OH) D | 4 month
  Considering the fifth day of the female monthly period (8-10 hours fasting), blood samples were taken from all participants following overnight fasting and within 48 hours before starting the test and just following 16-week exercise training and receiving vitamin D supplements.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alghadir AH, Gabr SA, Iqbal A. Concurrent effects of high-intensity interval training and vitamin D supplementation on bone metabolism among women diagnosed with osteoporosis: a randomized controlled trial. BMC Musculoskelet Disord. 2025 Apr 21;26(1):381. doi: 10.1186/s12891-025-08275-x. PMID 40259289